CLINICAL TRIAL: NCT04918355
Title: A Health System Wide Evaluation of Mandated Use and Clinical Decision Support Tools to Improve PDMP Utilization and Patient Outcomes
Brief Title: A Health System Wide Evaluation of Clinical Decision Support Tools to Improve PDMP Utilization and Patient Outcomes
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 19-1130; 20-0072 (Other Grant/Funding Number: Bureau of Justice Administration)
Record Dates: First submitted 2021-06-02; First posted 2021-06-08 (Actual); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Medication Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Compact Disks; Caffeine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Provider Group 1: no alert: Control group to enable tracking of temporal changes in prescribing. Providers will not see any alert.
- Provider Group 2: Mandated alert: Control group where providers will see a generic pop-up alert within the Electronic Health Record (EHR) whenever they initiate an opioid or benzodiazepine prescription without recording use of the PDMP. Patient risk factors are not assessed or presented in the alert. Providers in ambulatory clinics will not be assigned to this group. Alerts do not appear with patients with oncology or sickle cell diagnoses, or hospice discharge orders.
  Clinical Decision Support (CDS) alerts: CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
  Interventions: Other: Clinical Decision Support (CDS) alerts
- Provider Group 3: PDMP alert: Providers will see a pop-up alert within the Electronic Health Record (EHR) when they initiate an opioid or benzodiazepine prescription without recording use of the PDMP and patients have one or more positive risk factors based on past/current prescriptions received. Patient risk factors are assessed and presented in the alert. Risk factors included are numbers of active or recent opioid and benzodiazepine prescriptions, overlapping prescriptions, co-prescribing of benzodiazepines and opioids, and use of long-acting opioids in opioid naïve patients. Alerts do not appear with patients with oncology or sickle cell diagnoses, or hospice discharge orders. Clinical Decision Support (CDS) alerts: CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
  Interventions: Other: Clinical Decision Support (CDS) alerts
- Provider Group 4: PDMP + EHR alert: Providers will see a pop-up alert within the Electronic Health Record (EHR) when they initiate an opioid or benzodiazepine prescription without recording use of the PDMP and patients have one or more positive risk factors based on both prescriptions and other factors recorded in the patient's EHR. Patient risk factors are assessed and presented in the alert. Risk factors included the risks described in Group 3, along with a history of accidental opioid overdose, diagnosis of Opioid Use Disorder, multiple recent acute care incidents with opioid use, or high-risk psychiatric diagnoses. Alerts do not appear with patients with oncology or sickle cell diagnoses, or hospice discharge orders. Clinical Decision Support (CDS) alerts: CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
  Interventions: Other: Clinical Decision Support (CDS) alerts

INTERVENTIONS:
Other: Clinical Decision Support (CDS) alerts — CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
  Groups: Provider Group 2: Mandated alert; Provider Group 3: PDMP alert; Provider Group 4: PDMP + EHR alert

SUMMARY:
This is a study comparing three clinical decision support (CDS) tools to enhance care by easing health care provider review of the Colorado prescription drug monitoring program (PDMP) prior to prescribing opioids (pain medications often called narcotics) or benzodiazepines (sedatives or muscle relaxants). The tools screen information from the PDMP (a statewide database of filled controlled medication) and a patient's medical record to identify high-risk factors for overdose.

The tools only appear when relevant, are purely informational to facilitate an evidence-based practice (PDMP review) and do not dictate care or suggest changes in treatment.

The study will track how each of the tools are used and if providers use the PDMP. Secondary outcomes include if a controlled medication prescription was written and future opioid use by patients.

DETAILED DESCRIPTION:
Prior research by this team has shown that when emergency department (ED) prescribers are less likely to prescribe an opioid analgesic to patients at high-risk of overdose or misuse when they consult the Colorado Prescription Drug Monitoring Program (PDMP). Despite extensive work to reduce workflow and accessibility barriers to use of the PDMP, the majority of providers still do not use the PDMP when making prescription decisions. Clinical decision support (CDS) that is embedded in the Electronic Health Record (EHR) has promise as a tool to increase PDMP use, advance presentation of important PDMP data to providers and improve opioid safety without interrupting provider workflow.

This pragmatic, randomized study is designed to determine if:

* CDS tools that deliver focused, timely clinical information about high risk prescriptions to prescribers can improve use of the PDMP
* The use of focused CDS tools can decrease high-risk opioid prescribing
* The use of focused CDS tools is associated with better patient outcomes: decreasing high-risk, long-term, and aberrant opioid use

Specifically, we will test the hypotheses that:

1. Focused CDS tools will increase the percentage of high-risk prescriptions with a PDMP review, compared to the control group.
2. Focused CDS tools will decrease the percentage of high-risk controlled medication prescriptions, compared to the control group.

The alerts will fire for discharge prescriptions in all system emergency departments, inpatient facilities and ambulatory care facilities. Evaluation of patient risk as described below will be conducted automatically and for two of the three visible alerts, the provider will only see the alert if the patient meets high risk criteria. Providers in emergency departments and inpatient facilities will be randomized at the individual level, while providers selected to participate in the ambulatory setting will be randomized so that providers who prescribe at the same site or set of sets ( such as a series of primary care clinics staffed by an identifiable set of providers) will be in the arm to reduce contamination between the groups. Approximately 4000 providers will be included, based on historical staffing of UCHealth facilities.

Health encounters will be identified on the basis of an encounter with an enrolled provider. Automated risk assessment steps will be carried out on patients seen at included UCHealth facilities in the course of the year-long activation of the alerts. Based on historical patient counts, this is approximately 950,000 unique patients. Visit data will be retrospectively collected. This population is expected to be approximately 200,000 individuals.

The CDS only changes the provider interface with the PDMP and does not include any treatment recommendations or limit providers in any way from providing opioids or benzodiazepines if that is the best course of action in the provider's clinical judgement. Providers are not required to check the PDMP. The CDS is designed to enable access to the PDMP specifically focused on high risk prescriptions.

As the study implements an automated CDS, which is routinely introduced into clinical practice with no consent process, and does not make any treatment recommendations or requirements, it is being conducted at the provider level under a waiver of informed consent. Patient outcome determination will be conducted as secondary research, with patients to be included identified on the basis of their interaction with an enrolled health care provider. Only data collected as part of routine care will be collected to measure secondary outcomes. All patient data will be de-identified by the research team's Honest Broker and a de-identified data set provided for analysis.

ELIGIBILITY:
Two populations are included in the study description. Providers and the patients seen by those providers.

Providers are randomized to one of the four groups described previously.

Provider Inclusion Criteria:

* Licensed health care providers within the UCHealth system with a history (previous year) of prescribing opioids and/or benzodiazepines.

Provider Exclusion Criteria:

* Majority of prescribing is done at a facility outside the state of Colorado
* Provider specialty of oncology or pediatrics as recorded in the EHR
* Provider in an ambulatory clinic where a total of <50 opioid or benzodiazepine prescriptions were written in the year before study initiation

Patient Inclusion Criteria:

* Patient seen by a randomized provider within the UCHealth system who may receive an opioid prescription

Patient Exclusion Criteria:

* Less than 12 years of age or greater than 89 years of age at the time of the first study associated visit
* Active oncology or sickle cell diagnosis
* Active end of life care (defined as discharge to hospice or palliative care facility or specific palliative care orders in the medical record)

Ages: 12 Years to 89 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Provider population: Health care providers in Colorado who work in the University of Colorado Health (UCHealth) system.
  Patient population: Residents and visitors to the state of Colorado who seek healthcare within the UCHealth system.
Sampling Method: Non-Probability Sample
Enrollment: 3635 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Hoppe, DO, Principal Investigator — University of Colorado School of Medicine
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Providers prescribing at least 12 opioids + benzodiazepines in the prior year were selected for inclusion. Providers primarily working in inpatient and emergency department settings were randomized individually. Providers primarily working in an outpatient setting were randomized to assure providers working in the same clinics were in the same randomization arm. Enrollment numbers reported reflect the number of providers involved in the study as patients were not exposed to the intervention.
Pre-assignment Details: Outpatient providers were not included in the mandated arm as the provider group felt the alerts would be too interruptive.
Units Other Than Participants: Health care encounters
Groups:
- Provider Group 1: no Alert: Control group to enable tracking of temporal changes in prescribing. Providers will not see any alert. Providers were randomly assigned to an arm and any patients they saw as part of routine care were also considered to be in that arm during the encounter with the provider.
Period: Overall Study
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert
Started (health care providers were randomized prospectively and health care encounters were analyzed retrospectively.) | 1106; 22226 Health care encounters (Provider counts by clinical work settings: Emergency department- 141 (randomized at provider level); Inpatient- 325 (randomized at provider level); outpatient- 640 across 84 clinics (randomized at clinic level)) | 468; 17804 Health care encounters (Provider counts by clinical work settings: Emergency department- 142 (randomized at provider level); Inpatient- 326 (randomized at provider level); outpatient- 0 (setting would not allow this intervention)) | 973; 20840 Health care encounters (Provider counts by clinical work settings: Emergency department- 142 (randomized at provider level); Inpatient- 327 (randomized at provider level); outpatient- 504 across 82 clinics (randomized at clinic level)) | 1088; 27177 Health care encounters (Provider counts by clinical work settings: Emergency department- 141 (randomized at provider level); Inpatient- 324 (randomized at provider level); outpatient- 623 across 82 clinics (randomized at clinic level))
Completed (Providers were randomized into arms to be given a clinical decision support intervention. Upon retrospective health data extract several providers did not have any qualifying encounters in the system. Those counted as completed did have a qualifying health encounter.) | 609; 22226 Health care encounters | 276; 17804 Health care encounters | 535; 20840 Health care encounters | 664; 27177 Health care encounters
Not Completed | 497; 0 Health care encounters | 192; 0 Health care encounters | 438; 0 Health care encounters | 424; 0 Health care encounters
Not completed — no qualifying health encounter | 497 | 192 | 438 | 424

BASELINE CHARACTERISTICS:
Population: Baseline data was generated for patient characteristics of qualifying health care encounters. Randomized provider baseline data was not assessed.
Units Other Than Participants: health care encounter
Groups:
- Provider Group 3: PDMP Alert: Providers will see a pop-up alert within the EHR when they initiate an opioid or benzodiazepine prescription without recording use of the PDMP and patients have one or more positive risk factors based on past/current prescriptions received. Patient risk factors are assessed and presented in the alert. Risk factors included are numbers of active or recent opioid and benzodiazepine prescriptions, overlapping prescriptions, co-prescribing of benzodiazepines and opioids, and use of long-acting opioids in opioid naïve patients.
  Alerts are seen only once regardless of the number of positive risk factors and do not appear with patients with oncology or sickle cell diagnoses, or hospice discharge orders.
  Clinical Decision Support (CDS) alerts: CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
- Provider Group 4: PDMP + EHR Alert: Providers will see a pop-up alert within the EHR when they initiate an opioid or benzodiazepine prescription without recording use of the PDMP and patients have one or more positive risk factors based on both prescriptions and other factors recorded in the patient's Electronic Health Record. Patient risk factors are assessed and presented in the alert. Risk factors included the risks described as in Group 3, along with a history of accidental opioid overdose, diagnosis of Opioid Use Disorder, multiple recent acute care incidents with opioid use, or high risk psychiatric diagnoses.
  Alerts are seen only once regardless of the number of positive risk factors and do not appear with patients with oncology or sickle cell diagnoses, or hospice discharge orders.
  Clinical Decision Support (CDS) alerts: CDS alerts are pop-up boxes integrated into the EHR. Each alert provides patient specific information, a link to the PDMP, instructions on how to dismiss the alert, a link to study-specific educational website, and a comment field.
- Total: Total of all reporting groups
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert | Total
Number analyzed (Participants) | NA | NA | NA | NA | NA
Number analyzed (health care encounter) | 22226 | 17804 | 20840 | 27177 | 88047
Age, Customized [Count of Units; unit: health care encounter]
  Age: 18-64 years | 18410 | 15794 | 17327 | 22545 | 74076
  Age: 65 and over years | 3816 | 2010 | 3513 | 4632 | 13971
Sex: Female, Male [Count of Units; unit: health care encounter]
  Female | 14392 | 9739 | 13293 | 17166 | 54590
  Male | 7834 | 8065 | 7547 | 10011 | 33457
Ethnicity (NIH/OMB) [Count of Units; unit: health care encounter]
  Hispanic or Latino | 2899 | 3343 | 2510 | 3462 | 12214
  Not Hispanic or Latino | 19105 | 14236 | 18152 | 23354 | 74847
  Unknown or Not Reported | 222 | 225 | 178 | 361 | 986
Race (NIH/OMB) [Count of Units; unit: health care encounter]
  American Indian or Alaska Native | 104 | 97 | 129 | 171 | 501
  Asian | 37 | 76 | 39 | 53 | 205
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1065 | 1119 | 953 | 1023 | 4160
  White | 18225 | 13362 | 17386 | 22859 | 71832
  More than one race | 819 | 753 | 733 | 946 | 3251
  Unknown or Not Reported | 1976 | 2397 | 1600 | 2125 | 8098
Region of Enrollment [Number; unit: health care encounter]
  United States | 22226 | 17804 | 20840 | 27177 | 88047
Medication type triggering alert [Count of Units; unit: health care encounter]
  benzodiazepine | 6088 | 1946 | 6814 | 8285 | 23133
  opioid | 15545 | 15655 | 13333 | 18345 | 62878
  benzodiazepine and opioid | 593 | 203 | 693 | 547 | 2036

OUTCOME MEASURES:

1. Primary Outcome: Percentage of PDMP Checks Conducted During High-risk Prescriptions
Description: Differences between groups in the percentage of opioid or benzodiazepine prescriptions with one or more high risk prescribing criteria for whom the health care provider consults the Prescription Drug Monitoring Program (PDMP) prior to signing, in line with prescribing best practices.
Time Frame: Total over the course of one year
Population: Health encounter with a high-risk prescription written
Measure: Count of Units; unit: health care encounters
Units Other Than Participants: health care encounters
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (health care encounters) | 22226 | 7622 | 20840 | 27177
health care encounters | 8187 | 6322 | 13360 | 23328

2. Secondary Outcome: Percentage of High-risk Controlled Medication Prescriptions Abandoned
Description: Differences between groups in the percentage of encounters with one or more high risk prescribing criteria where the provider does not sign a prescription for an opioid after initiating the prescription and seeing the intervention reminding the provider to check the PDMP (CDS tool fires).
Time Frame: Total over the course of one year
Population: Health care encounters with a high risk prescribed medication that triggered clinical decision support alert.
Measure: Count of Units; unit: health care encounters
Units Other Than Participants: health care encounters
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (health care encounters) | 16138 | 6522 | 14026 | 18892
health care encounters | 538 | 605 | 768 | 1314

3. Secondary Outcome: Long Term Opioid Use
Description: Number of encounters where the patient experiences long term or aberrant opioid use (combined metric).
Time Frame: Total over the course of one year
Population: high risk opioid prescription medical visits for patients seen again in the hospital system
Measure: Count of Units; unit: health care encounters
Units Other Than Participants: health care encounters
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert
Number analyzed (Participants) | NA | NA | NA | NA
Number analyzed (health care encounters) | 16138 | 18892 | 6522 | 14026
health care encounters
  chronic opioid use | 3,233 | 5,565 | 573 | 2,414
  aberrant opioid use | 503 | 731 | 310 | 433

ADVERSE EVENTS:
Time Frame: Approximately 15 minutes, during health encounter
Description: Adverse evens were extracted from the healthcare encounters. The number at risk represents the total number of healthcare encounters analyzed for adverse events.
  Providers were not assessed for deaths or adverse events as the intervention is an electronic display of data within the providers' typical workflow within the electronic health record system. Patient outcomes were considered the outcome of routine health care, not of the intervention being studied.
Arm/Group | Provider Group 1: no Alert | Provider Group 2: Mandated Alert | Provider Group 3: PDMP Alert | Provider Group 4: PDMP + EHR Alert
All-Cause Mortality (participants affected / at risk) | 0/22226 | 0/17804 | 0/20840 | 0/27177
Serious Adverse Events (participants affected / at risk) | 0/22226 | 0/17804 | 0/20840 | 0/27177
Other Adverse Events (participants affected / at risk) | 0/22226 | 0/17804 | 0/20840 | 0/27177

LIMITATIONS AND CAVEATS:
Providers were randomized, health visits in which an opioid or benzodiazepine was prescribed were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04918355/Prot_SAP_000.pdf